CLINICAL TRIAL: NCT01648608
Title: Study to Assessment the Efficacy and Safety of Joint TAC and Exemestane as Neoadjuvant Chemotherapy in the Postmenopausal Women With Operable Breast Cancer
Brief Title: Efficacy and Safety of TAC and Exemestane as Neoadjuvant Chemotherapy in the Postmenopausal Women With Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Zhang jin, Professor, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENBC
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exemestane (Experimental): Exemestane for neoadjuvant chemotherapy
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — Exemestane for neoadjuvant chemotherapy

SUMMARY:
Select the postmenopausal patients with breast cancer who is confirmed by core needle biopsy and at the clinical stage T2-4N0-2M0.Treat them with 4 cycles of TAC as neoadjuvant chemotherapy (Docetaxel was 75mg/m2, the EPI 60mg/m2 and the CTX 600mg/m2,21day/cycle).At the same time give daily oral exemestane 25mg for 12 weeks.Then assess the efficacy and safety of TAC and Exemestane.

DETAILED DESCRIPTION:
The investigators select the postmenopausal patients with breast cancer who is confirmed by core needle biopsy and at the clinical stage T2-4N0-2M0.Treat them with 4 cycles of TAC as neoadjuvant chemotherapy (Docetaxel was 75mg/m2, the EPI 60mg/m2 and the CTX 600mg/m2,21day/cycle).At the same time give daily oral exemestane 25mg for 12 weeks.Then assess the efficacy and safety of TAC and Exemestane.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky ≥ 70
2. Provision of informed consent
3. Pathological confirmation of invasive ductal carcinoma and estrogen receptor is positive
4. Tumor stage(TNM):T2-4bN0-3M0
5. Premenopausal woman
6. Not previously received treatment with bisphosphonate
7. Laboratory criteria:

   * PLT ≥ 100*109/L
   * WBC ≥ 4000/mm3
   * HGB ≥ 10g/dl
   * GOT,GPT,ALP ≤ 2*ULN
   * TBIL,DBIL,CCr ≤ 1.5*ULN

Exclusion Criteria:

1. Pregnant or lactation woman
2. History of organ transplantation
3. With mental disease
4. With severe infection or active gastrointestinal ulcers
5. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
6. Disease-free period of other malignant tumor is less than 5 years(except cured basal cell skin cancer and cervical carcinoma in situ)
7. With heart disease
8. Experimental drug allergy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
therapeutic assessment | 6 months
  therapeutic assessment

SECONDARY OUTCOMES:
Adverse reactions and disease-free survival | 2 years
  Adverse reactions and disease-free survival

OTHER OUTCOMES:
Recurrence or death | 5 years
  Recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: jin Zhang, Professor, Study Chair — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China